CLINICAL TRIAL: NCT04665843
Title: A Phase II, Randomized, Double Blind Study of Atezolizumab Plus Tiragolumab and Atezolizumab Plus Placebo as First-Line Treatment in Patients With Recurrent/Metastatic PD-L1 Positive Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study of Atezolizumab Plus Tiragolumab and Atezolizumab Plus Placebo as First-Line Treatment in Participants With Recurrent/Metastatic PD-L1 Positive Squamous Cell Carcinoma of the Head and Neck
Acronym: SKYSCRAPER-09
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BO42533; 2020-002852-19 (EudraCT Number)
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — atezolizumab; Tiragolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Tiragolumab (Experimental): Participants will receive atezolizumab followed by tiragolumab every three weeks (Q3W) on Day 1 of each 21-day cycle.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Atezolizumab + Placebo (Placebo Comparator): Participants will receive atezolizumab followed by placebo Q3W on Day 1 of each 21-day cycle.
  Interventions: Drug: Atezolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab at a fixed dose of 1200 mg will be administered by intravenous (IV) infusion Q3W on Day 1 of each 21-day cycle.
  Other Names: Tecentriq; RO5541267
Drug: Tiragolumab — Tiragolumab at a fixed dose of 600 mg will be administered by IV infusion Q3W on Day 1 of each 21-day cycle.
  Other Names: RO7092284
  Arms: Atezolizumab + Tiragolumab
Drug: Placebo — Placebo will be administered by IV infusion Q3W on Day 1 of each 21-day cycle.
  Arms: Atezolizumab + Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of atezolizumab plus tiragolumab and atezolizumab plus placebo as first-line (1L) treatment in recurrent/metastatic PD-L1-positive squamous cell carcinoma of the head and neck (SCCHN) on the basis of confirmed objective response rate. In addition, safety, pharmacokinetics, immunogenicity of atezolizumab and tiragolumab will be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed recurrent/metastatic SCCHN involving the oropharynx, oral cavity, larynx, or hypopharynx, that is considered incurable by local therapies
* Known results from human papillomavirus (HPV) status test for oropharyngeal carcinoma
* No prior systemic therapy for metastatic and/or recurrent SCCHN
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Tumor PD-L1 expression as determined by PD-L1 immunohistochemistry assay
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy >=12 weeks

Key Exclusion Criteria:

* Disease suitable for local therapy with curative intent
* Progressive or recurrent disease within 6 months of the last dose of curative intent systemic treatment for locally advanced SCCHN
* Rapidly progressing disease in the opinion of the treating investigator
* Grade >=2 unresolved toxicity related to surgery or other prior therapies
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* History of additional malignancy other than SCCHN within 5 years prior to randomization
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-TIGIT, anti-PD-L1, and anti-PD-1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents or systemic immunosuppressive medication
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) | Up to approximately 43 months

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 43 months
Progression-Free Survival (PFS) | Up to approximately 43 months
Overall Survival (OS) | Up to approximately 43 months
Progression-Free Survival Rate at 6 Months | Month 6
Overall Survival Rate at 6 Months and 12 Months | Month 6, Month 12
Time to Confirmed Deterioration (TTCD) in Patient-Reported Physical Functioning | Up to approximately 43 months
Percentage of Participants With Adverse Events (AEs) | Up to approximately 43 months
Minimum Serum Concentration (Cmin) of Atezolizumab | Predose and 30 minutes postdose on Day 1 of Cycle 1 (each cycle is 21 days), predose on Day 1 of Cycles 2, 3, 4, 8, 12, 16 and at treatment discontinuation visit up to approximately 43 months
Maximum Serum Concentration (Cmax) of Atezolizumab | Predose and 30 minutes postdose on Day 1 of Cycle 1 (each cycle is 21 days), predose on Day 1 of Cycles 2, 3, 4, 8, 12, 16 and at treatment discontinuation visit up to approximately 43 months
Cmin of Tiragolumab | Predose and 30 minutes postdose on Day 1 of Cycle 1 (each cycle is 21 days), predose on Day 1 of Cycles 2, 3, 4, 8, 12, 16 and at treatment discontinuation visit up to approximately 43 months
Cmax of Tiragolumab | Predose and 30 minutes postdose on Day 1 of Cycle 1 (each cycle is 21 days), predose on Day 1 of Cycles 2, 3, 4, 8, 12, 16 and at treatment discontinuation visit up to approximately 43 months
Number of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab | From baseline up to approximately 43 months
Number of Participants With ADAs to Tiragolumab | From baseline up to approximately 43 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (47):
- United States (7):
  - Moores Cancer Center at UC San Diego Health, La Jolla, California
  - UCLA, Los Angeles, California
  - SCRI Florida Cancer Specialists PAN, Tallahassee, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Czechia (3):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice v Motole, Prague
- France (6):
  - CHU Bordeaux, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Leon Berard, Lyon
  - Institut régional du Cancer Montpellier, Montpellier
  - Institut Curie, Paris
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
- Greece (4):
  - Anticancer Hospital Ag Savas, Athens
  - Attiko Hospital University of Athens, Athens
  - Periph. University General Hospital of Heraklion Crete, Heraklion
  - Euromedical General Clinic of Thessaloniki, Thessaloniki
- Hungary (3):
  - Gy?r-Moson-Sopron Vármegyei Petz Aladár Egyetemi Oktató Kórház, Gy?r
  - Bacs-Kiskun Megyei Korhaz, SZTE AOK Oktato Korhaza, Onkoradiologiai Kozpont, Kecskemét
  - Pécsi Tudományegyetem, Pécs
- Italy (3):
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
- Auckland City Hospital, Cancer and Blood Research, Auckland, New Zealand
- Poland (5):
  - Beskidzkie Centrum Onkologii- Szpital Miejski, Bielsko-Biala
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Centrum Terapii Wspolczesnej J.M.Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Centrum Onkologii Ziemi Lubelskiej Im. ?W. Jana Z Dukli, Lublin
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Zhongzheng Dist.
- Thailand (2):
  - Ramathibodi Hospital, Bangkok
  - Songklanagarind Hospital, Songkhla
- United Kingdom (4):
  - Velindre Cancer Centre, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing